CLINICAL TRIAL: NCT00356993
Title: The STOP (Stop Smoking Therapy for Ontario Patients) Study: The Effectiveness of Nicotine Replacement Therapy in Ontario Smokers.
Brief Title: Phase I Study: Stop Smoking Therapy for Ontario Patients (STOP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Peter Selby, Chief, Addictions Program, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81/2005
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Results first posted 2019-05-02 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Smoking
Keywords: nicotine replacement therapy; smoking cessation
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Nicotine Replacement Therapy; Tobacco Use Cessation Devices; Nicotine Chewing Gum; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NRT + Behavioural Support (Experimental): Nicotine Replacement Therapy plus Behavioural Intervention
  Interventions: Drug: Nicotine Replacement Therapy; Behavioral: behavioural intervention

INTERVENTIONS:
Drug: Nicotine Replacement Therapy — transdermal nicotine patch, nicotine gum, nicotine inhaler, nicotine lozenge
  Other Names: transdermal nicotine patch; nicotine gum; nicotine inhaler; nicotine lozenge
Behavioral: behavioural intervention — Smoking cessation counselling, relapse prevention strategies

SUMMARY:
20% of Ontarians smoke. There was a decline in smoking prevalence from 1995 but it has remained unchanged since 2002. This rate of smoking cessation has not kept up with the rest of Canada. A new strategy is necessary to increase the number of smokers making quit attempts and to increase the odds of quitting long term.The goal of this study is to evaluate the methods and effectiveness of providing nicotine replacement (NRT) to Ontario smokers. The study will develop an evidence-based protocol for providing NRT, provide faculty development on combining pharmacotherapy with behavioural interventions and will provide an evaluation framework to inform future coverage models.

DETAILED DESCRIPTION:
According to the US Surgeon General's Report (1988), there are immediate, intermediate and long-term benefits to health from quitting smoking. For example, there is a 50% reduction in coronary heart disease risk in 12 months and the risk of a stroke is reduced to that of a nonsmoker 5-15 years after quitting. (US Surgeon General's Report, 1990, p.vi). In a systematic assessment of the value of clinical preventive services recommended by the US Preventive Services Task Force, smoking cessation treatment for adults was one of the highest-ranked services in terms of its cost effectiveness and its potential to reduce the burden of disease. Most smoking cessation interventions cost less per year of life saved than most widely accepted medical practices. For example, cost-effectiveness analysis of the implementation of the Agency for Healthcare Research and Quality (AHRQ) guidelines show costs of $4,113 per life-year saved, in 2001 prices compared to annual mammography for women aged 40 to 49 years, which costs $71,751 in 2001 prices, and hypertension screening for men aged 40 years, which costs $27,117 in 2001 prices. Therefore, smoking cessation services have been referred to as the "gold standard" for comparing the cost effectiveness of other healthcare interventions. Although some studies have shown high costs from increased healthcare utilization in the first year after quitting smoking due to illness (Martinson, 2003), most studies demonstrate that smokers who quit eventually have significantly lower healthcare utilization than continuing smokers (Fishman, 2003; Warner, 2003) Thus, for healthcare organizations such as the Ontario Health Insurance Plan, implementing smoking cessation services will likely result in a relatively quick return on investment. Both the intensity and duration of behavioural interventions are associated with sustained remission in smoking. The addition of pharmacotherapy doubles the odds of quitting successfully. However, many smokers face barriers in accessing pharmacotherapy. The provision of free pharmacotherapy has the potential to help a substantial number of smokers to quit. A study by Curry et al, 1998, evaluated smokers who were willing to sign up for a cessation-support program under various degrees of coverage for either the program or nicotine replacement therapy (NRT). 10% of Smokers with full coverage were likely to attempt to quit as opposed to 2.5% with partial coverage. Therefore, the USHHS guidelines call for the coverage of these medications. Research has shown that coverage for tobacco dependence treatments can enhance not only the rate of quit attempts but also long-term abstinence for smokers (Levy & Friend, 2002; Schauffler, McMenamin, Olson, Boyce-Smith, Rideout, & Kamil, 2001). On average, the odds ratio of quitting at one year was 1.6 for those given free NRT. Therefore, some insurers, both public and private, reimburse patients for stop smoking medications. However, a study by Boyle et al 2002, found that simply including the medication in an insurance plan did not increase quit rates or utilization of medications. Adequate precautions must be taken to ensure that free pharmacotherapy is distributed in conjunction with behavioural interventions to be successful and to be used by those smokers most likely to benefit from pharmacotherapy.Pharmacotherapy can be very expensive if provided to all smokers. However, not all smokers want to quit or require medications to quit (McDonald, 2003). Most smokers use about 2-3 weeks of pharmacotherapy when not combined with behavioural interventions (Pierce, 2002). About 0.05% of smokers looking to quit will seek specialized care. Moreover, if we assume that 70% of current tobacco users (Approximately 1.6 million) in Ontario will try to quit in a given year and that 10% ( i.e. 169,000) of these individuals would qualify for and seek reimbursement for 10 weeks of therapy at $30/week, then the total estimated cost will be about $50 million! This is clearly not fundable and therefore a comprehensive strategy combined with some rational use of pharmacotherapy is necessary.Hypothesis:

The provision of free NRT will increase long-term quit rates (>/= 6 months) in Ontario smokers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be Ontario residents
* Older than or equal to 18 years of age
* Current daily smokers who smoke >10 cigarettes per day
* Smoked more than 100 cigarettes in their lifetime

Exclusion Criteria:

* Current treatment with Varenicline
* Allergic to adhesive
* Intolerant to Nicotine Replacement Therapy
* Medical contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6009 (Actual)
Dates: Start 2005-10; Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Selby, MD, MHSc, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research
- See also: click for more information on the study: The STOP (Stop Smoking Therapy for Ontario Patients) Study: The Effectiveness of Nicotine Replacement Therapy in Ontario Smokers. — https://www.nicotinedependenceclinic.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NRT + Behavioural Support
Started | 6009
Completed | 2088
Not Completed | 3921

BASELINE CHARACTERISTICS:
Arm/Group | NRT + Behavioural Support
Number analyzed (Participants) | 6009
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: missing information for 9 participants
  years
    number analyzed (Participants) | 6000
    (all) | 47.6 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: missing data n=9
  Participants
    number analyzed (Participants) | 6000
    Female | 3201
    Male | 2799
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Cigarettes per day (cpd) [Count of Participants; unit: Participants] — Population: missing information for 3921 participants
  Participants
    number analyzed (Participants) | 2088
    1-9 cigarettes | 6
    10-14 cigarettes | 358
    15-19 cigarettes | 337
    20-24 cigarettes | 493
    25+ cigarettes | 888
    No response | 6
Age started to smoke daily [Mean (Standard Deviation); unit: years] | 17.3 (4.8)
Age first smoked [Mean (Standard Deviation); unit: years] | 14.2 (5.1)
Number of Quit Attempts in past year [Count of Participants; unit: Participants] — Population: Missing data n= 245
  Participants
    number analyzed (Participants) | 5764
    0 quit attempt | 3058
    1 quit attempt | 2328
    2 quit attempts | 378
Importance of Quitting [Count of Participants; unit: Participants] — A scale of 1 to 10 , where 10 means the most important thing and 1 is the least important thing to do. Population: missing data n=29
  Participants
    number analyzed (Participants) | 5980
    1-least important thing to do | 22
    2 | 10
    3 | 13
    4 | 14
    5 | 70
    6 | 66
    7 | 217
    8 | 797
    9 | 802
    10- the most important thing to do | 3969
Confidence to Quit Smoking [Count of Participants; unit: Participants] — Scale of 1 to 10
  1 -very little confidence 10- very confident that you can quit Population: missing data n=47
  Participants
    number analyzed (Participants) | 5962
    1- very little confidence | 66
    2 | 95
    3 | 138
    4 | 170
    5 | 870
    6 | 506
    7 | 859
    8 | 1373
    9 | 591
    10 -very confident | 1294
Diagnosed with a psychiatric disorder [Count of Participants; unit: Participants]
  Yes- diagnosed with a psychiatric disorder | 2447
  not diagnosed or missing data | 3562
highest level of education attained [Count of Participants; unit: Participants] — Population: missing data n=76
  Participants
    number analyzed (Participants) | 5933
    some primary school | 94
    Primary school | 164
    some high school | 1235
    high school diploma | 1369
    some college | 853
    College diploma | 1269
    Some university | 404
    University degree | 545

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants Not Smoking
Description: 7-day point prevalence of abstinence at 6 months post treatment
Time Frame: 6 months post treatment
Population: Not every participant completed the 6mo and 12mo follow-up surveys
Measure: Count of Participants; unit: Participants
Arm/Group | NRT + Behavioural Support
Number analyzed (Participants) | 2088
Participants | 766

2. Secondary Outcome: Count of Participants Not Smoking
Description: 7-day point prevalence of abstinence at 12 months post treatment
Time Frame: 12 months post treatment
Population: Not every participant completed the 12mo follow-up surveys
Measure: Count of Participants; unit: Participants
Arm/Group | NRT + Behavioural Support
Number analyzed (Participants) | 387
Participants | 147

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | NRT + Behavioural Support
All-Cause Mortality (participants affected / at risk) | 0/6009
Serious Adverse Events (participants affected / at risk) | 0/6009
Other Adverse Events (participants affected / at risk) | 0/6009

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2006-03-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT00356993/Prot_000.pdf